CLINICAL TRIAL: NCT07142265
Title: Evaluation of 1-Year Clinical Outcomes With Early Inclisiran Initiation in Post-MI Patients
Acronym: STREAMLINE
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839D1RU01
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; NIS; inclisiran
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI/Non-STEMI: Patients with inclisiran initiation in 14 ± 5 days after STEMI/non-STEMI

SUMMARY:
Evaluation of clinical outcomes during 12 months after inclisiran initiation in patients after STEMI/non-STEMI in real-world settings in Russia. It is also planned to study the therapy effect on the lipid profile characteristics, its safety, the state of atherosclerotic plaques according to carotid ultrasound, the frequency of hospitalizations and the need for intensive follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders
* Myocardial Infarction diagnosis
* Dyslipidemia diagnosis
* The first injection of inclisiran no later than 14 ± 5 days after the STEMI/non-STEMI
* LDL-C > 5 mmol/L (statin-naive patients) or LDL-C > 2.5 mmol/L (on the basis of statin MTD) at the time of hospitalization or no target LDL-C level (> 1.4 mmol/L or no LDL-C level decrease by 50% on statin MTD + ezetimibe)
* Signed Informed Consent Form (ICF)

Exclusion Criteria:

* Severe oncological and somatic diseases with system and organ failure*
* Competing diseases that caused emergency hospitalization (pulmonary thromboembolism, aortic dissection)
* History of therapy with PCSK9 inhibitors
* Active inflammatory liver disease or the levels of AST, ALT > 3 times, or total bilirubin > 2 times higher than the upper limit of norm
* Any other MACE in the anamnesis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with inclisiran initiation in 14 ± 5 days after STEMI/non-STEMI. Index event is a first diagnosed STEMI/non-STEMI.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Atherosclerotic Cardiovascular Disease (ASCVD) events registered within 12 months after inclisiran initiation in addition to basic therapy | 12 months
  Number of patients with Atherosclerotic Cardiovascular Disease (ASCVD) events (cardiac death, nonfatal MI, nonfatal ischemic stroke, and hospitalization for unstable angina) registered within 12 months after the start of inclisiran therapy prescribed in addition to basic LLT

SECONDARY OUTCOMES:
Change and absolute change in lipid profile parameters | Baseline, month 3, month 9, month 12
  Change and absolute change in lipid profile parameters (total cholesterol, LDL-C, HDL-C, non-HDL-C, triglycerides, lipoprotein (a)) at 3, 9, and 12 months
Change and absolute change in lipid profile parameters in patients subgroups | Baseline, month 3, month 9, month 12
  Change and absolute change in lipid profile parameters at 3, 9, and 12 months in each of the 3 groups of patients identified on the basis of therapy and LDL-C level at admission:
  1. Patients who have not previously received statins, with LDL-C level > 5 mmol/L;
  2. Patients receiving MTD statin therapy with LDL-C level of > 2.5 mmol/L;
  3. Patients receiving MTD statin therapy + ezetimibe who not at LDL-C target (> 1.4 mmol/L) or did not achieve a 50% reduction in LDL-C level
Change in LDL-C level | Baseline, Day 28
  Change in LDL-C level at Day 28 from baseline
The proportion of patients who maintain the target LDL-C level | Month 3, Month 12
  The proportion of patients who maintain the target LDL-C level achieved after 3 months throughout the study period (12 months)
The proportion of patients who achieved the target LDL-C level of < 1.4 mmol/L | Day 28 , Month 12
  The proportion of patients who achieved the target LDL-C level of < 1.4 mmol/L at Day 28 and at 12 months
The proportion of patients with progression and regression/no changes in atherosclerotic plaque | Baseline, Month 12
  The proportion of patients with progression and regression/no changes in atherosclerotic plaque determined on the basis of changes in its maximum height (mm) by carotid ultrasound at 12 months compared to 3-5 days after ACS (Acute Coronary Syndrome)
Number (%) of patients who achieved the target LDL-C level of < 1.4 mmol/L and with change in the maximum plaque height (mm) | 12 months
  The correlation between the achievement of the target LDL-C level of < 1.4 mmol/L and a change in the maximum plaque height (mm) is going to be measured.
Total number of patients with adverse events (AE) in general, treatment-emergent AE (TEAEs), and serious adverse events (SAE) | Month 3, Month 9, Month 12
  Total number of patients with adverse events (AE) in general, treatment-emergent AE (TEAEs), and serious adverse events (SAE) at 3, 9, and 12 months
The number of patients who discontinued inclisiran therapy due to AEs | Month 3, Moth 9, Month 12
  The number of patients who discontinued inclisiran therapy due to AEs at 3, 9, and 12 months
The number of patients re-hospitalized for CV events during the year | 12 months
  The number of patients re-hospitalized for cardiovascular (CV) events during the year
The number of patients re-hospitalized during the year for scheduled and unscheduled revascularization | 12 months
  The number of patients re-hospitalized during the year for scheduled and unscheduled revascularization
Number of patients who sought emergency care after the baseline visit | 12 months
  Number of patients who sought emergency care after the baseline visit
The number of patients placed under dispensary observation | 12 months
  The number of patients placed under dispensary observation
Number of days from the date of hospital discharge to place under dispensary observation | 12 months
  Number of days from the date of hospital discharge to place under dispensary observation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Russia (7):
  - Novartis Investigative Site, Cheboksary
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ulan-Ude

IPD SHARING:
Plan to Share IPD: No